CLINICAL TRIAL: NCT00501371
Title: Double-Blind, Randomized, Placebo-Controlled Study to Investigate the Efficacy and Safety of MCS in Treating Lower Urinary Tract Symptoms Suggestive of Benign Prostatic Hyperplasia
Brief Title: MCS in Treating Lower Urinary Tract Symptoms (LUTS) Suggestive of Benign Prostatic Hyperplasia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated for re-design. A new IND study (US FDA, July 2009) will be conducted in US and Taiwan. Termination not related to safety concerns.
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCS for BPH-LUTS
Record Dates: First submitted 2007-07-10; First posted 2007-07-16 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; MCS; Lower Urinary Tract Symptoms; International prostate symptom score; Voiding; Alpha-blockers
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCS (Active Comparator): Group A: MCS 30 mg/day for 12 weeks
  Interventions: Drug: MCS
- Placebo (Placebo Comparator): Placebo, 2 capsules per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCS — soft-gel capsule, 15 mg/cap., Qd, 12 weeks
  Other Names: MUS
  Arms: MCS
Drug: Placebo — soft-gel capsule, Qd, 12 weeks
  Other Names: MUS
  Arms: Placebo

SUMMARY:
Phase III, Randomized, double-blind, parallel placebo-controlled study. Two arms: MCS (30mg/day) vs. placebo.

Subproject MCS-2: alpha-blocker naïve subjects

Subproject MCS-3: subjects responding poorly to alpha-blocker

DETAILED DESCRIPTION:
For MCS-2 This is a double-blind, randomized, placebo-controlled, parallel study where eligible male subjects (age 40, N=188), after a two-week washout period, will be randomized at 1:1 ratio to receive either MCS 30 mg/day or placebo for 12 weeks.

Group A: MCS 30 mg/day for 12 weeks Group B: placebo for 12 weeks

Subjects are limited to those who are currently not being treated medically for BPH or LUTS with alpha-blockers, anti-cholinergics, 5-alpha reductase inhibitors, or hormonal therapeutic agents. For each treatment arm, about 85 subjects eligible for final per protocol analysis will be recruited. Concerning an expected dropout rate of 10%, 188 subjects in total will be recruited onto the study.

For MCS-3 This is a double-blind, randomized, placebo-controlled, add-on, parallel study where eligible male subjects (age 40, N=242), after a two-week washout period, will be randomized at 1:1 ratio to receive either MCS 30 mg/day plus alpha-blocker or placebo plus alpha-blocker for 12 weeks.

Group A: alpha-blocker plus MCS 30 mg/day Group B: alpha-blocker plus placebo

Subjects are limited to those who are currently not being treated medically for BPH or LUTS with anti-cholinergics, 5-alpha reductase inhibitors, or hormonal therapeutic agents. For each treatment arm, about 220 subjects eligible for final per protocol analysis will be recruited. Concerning an expected dropout rate of 10%, 242 subjects in total will be recruited onto the study.

All participating subjects will be advised to maintain a normal diet as they do before joining the study. However, participating subjects are advised to refrain from extra source of carotenoids supplementation and MCS extracts made into a capsule, soft gel, or crude granule extracts.

ELIGIBILITY:
Inclusion criteria for subproject MCS-2

* Age ≧ 40 years old.
* Not being treated for BPH or LUTS with Alpha-blocker, anti-cholinergics, 5-alpha reductase inhibitors, or hormonal agents.
* PSA≦4 ng/ml within 4 weeks of V1 and no pathologically-proven prostate cancer.
* No known malignancy, except cancers without signs of recurrence for > 5 years and no need for further anti-cancer treatment.
* AST/ALT≦3X UNL.
* creatinine≦3X UNL.
* Subjects who sign the informed consent form.

Exclusion criteria

* Subjects' LUTS are not BPH-related but are associated with such conditions as urethral stricture, prostatitis, neurogenic bladder, or pelvic treatment procedures.
* Have been treated with pelvis irradiation or pelvic surgery.
* Plan to undergo any invasive procedures within the study period, such as, prostate surgery, prostate biopsy, cystourethroscopy, pelvic surgery, laparotomy, or any procedures needing urethral catheterization.
* Participating in another investigational agent study in the past 12 weeks or are going to do so during the study period.
* Active infection or inflammation.
* Considered ineligible by the investigators.

Inclusion criteria for subproject MCS-3

* Age≧40 years old.
* The alpha-blocker dosage used should be as high as subjects can tolerate.
* No known malignancy, except cancers without signs of recurrence for > 5 years and no need for further anti-cancer treatment.
* PSA≦10.0 ng/ml without pathologically-proven prostate cancer or other cancers. Prostate biopsy is mandatory > 12 weeks before screening, if PSA is≧4 ng/ml to rule out prostate cancer.
* AST/ALT≦3X UNL.
* Creatinine≦3X UNL.
* Subjects who sign the informed consent form.

Exclusion criteria

* Subjects' LUTS are not BPH-related but associated with such conditions as urethral stricture, prostatitis, neurogenic bladder, or pelvic treatment procedures.
* Subjects who have been treated with pelvis irradiation or pelvic surgery.
* PSA > 10.0 ng/ml, abnormal DRE of the prostate or any suspicion of prostate malignancy. However, those who have a negative prostate biopsy are allowed.
* Active infection or inflammation.
* Considered ineligible by the investigators.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
MCS-2: To compare changes in I-PSS points after 12 weeks of MCS or placebo supplementation. | 12 weeks
MCS-3: To compare the percentage of subjects who achieve an I-PSS reduction by 4 or more points from baseline at 12 weeks between the MCS and the placebo arms. | 12 weeks

SECONDARY OUTCOMES:
To evaluate the general safety and tolerability. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Chang Gung Memorial Hospital, Chiayi City
  - Chung-Ho Memorial Hospital,Kaohsiung Medical University, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei